CLINICAL TRIAL: NCT02417376
Title: Effect of Nonsurgical Periodontal Treatment on Systemic Risk Markers of Cardiovascular Disease Clinically and Biochemically: A Randomized Trial
Brief Title: Changes in the Risk Factors of Coronary Heart Disease Observed After Scaling and Root Planing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government College of Dentistry, Indore (Other)
Responsible Party: Principal Investigator, Dr DIVYA SINGH HADA, Post-graduate Student, Government College of Dentistry, Indore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCD-010/55/2013
Record Dates: First submitted 2015-04-04; First posted 2015-04-15 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Coronary Heart Disease; Periodontitis
Keywords: Coronary heart disease; Periodontitis; C-reactive protein; Blood pressure
MeSH Terms: conditions — Coronary Disease; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Active Comparator): Periodontal intervention in the form of scaling and root planing by:
  1. ultrasonic piezoelectric scaler (frequency of 28-36 KHz) and
  2. gracey curets (set of 7 instruments number 1-14) to remove supra and subgingival calculus on teeth, is completed in two appointments of 45 to 60 min, within 24 hours
  Interventions: Device: piezoelectric ultrasonic scaler (frequency of 28-36 KHz); Device: Gracey curettes
- Control (No Intervention): No periodontal intervention in any form.

INTERVENTIONS:
Device: piezoelectric ultrasonic scaler (frequency of 28-36 KHz) — Periodontal treatment in the form of scaling and root planing (SRP) is provided to the patients assigned to the experimental group, after baseline examination. Scaling is performed using piezoelectric ultrasonic scaler (frequency of 28-36 KHz) and root planing is performed using area specific Gracey curettes (set of 7 instruments number #1-14). SRP is completed in two appointments of 45 min to 1 hour, within 24 hours period.
  Arms: Experimental
Device: Gracey curettes — set of 7 instruments number #1-14
  Arms: Experimental

SUMMARY:
The purpose of this study is to determine whether scaling and root planing as a periodontal intervention helps in improving the overall health of patients suffering from coronary heart disease.

DETAILED DESCRIPTION:
This study is a randomized, outcome assessor blinded, parallel group, trial to evaluate the effect of non surgical periodontal treatment in the form of scaling and root planing on coronary heart disease patients. 70 clinically defined coronary heart disease (CHD) patients with mild to moderate periodontitis, were allocated into two groups- experimental and control, in a ratio of 1:1. Scaling and root planing was provided as the intervention to the experimental group. To the control group no periodontal intervention in any form was provided. The primary outcome assessed is the changes in C-reactive protein level at baseline and after 1, 3, and 6 months of periodontal intervention. The secondary outcomes assessed are lipid profile, white blood cells (WBC) profile, and blood pressure (systolic and diastolic) at baseline and after 1, 3, and 6 months of periodontal intervention. Periodontal parameters including plaque index (PI), gingival index (GI), bleeding on probing (BOP), periodontal probing depth (PPD), and clinical attachment loss (CAL) is also assessed at baseline and after 6 months. All these parameters were also compared with their corresponding values in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Male and female > 35 yrs of age
* Clinically diagnosed stable CHD cases
* No other systemic disease
* Non-smoker
* Advanced chronic gingivitis and mild to moderate chronic periodontitis (≥ 4 teeth with probing depth ≤ 5 mm) and ≥ 14 teeth (excluding third molars)
* No periodontal therapy in the last 12 months.

Exclusion Criteria:

* Not fulfilling criteria of the defined CHD case
* Present smoker
* Pregnant or lactating females
* Suffering from any other systemic disease like diabetes
* Taking systemic antibiotic therapy in the last 3 months
* Advanced chronic periodontitis (probing depth > 5mm) and <14 teeth (excluding third molars)
* Received any periodontal therapy within last 12 months.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Divya S. Hada, PG Student, Principal Investigator — Government College of Dentistry

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] D'Aiuto F, Parkar M, Nibali L, Suvan J, Lessem J, Tonetti MS. Periodontal infections cause changes in traditional and novel cardiovascular risk factors: results from a randomized controlled clinical trial. Am Heart J. 2006 May;151(5):977-84. doi: 10.1016/j.ahj.2005.06.018. PMID 16644317
- [Result] Bokhari SA, Khan AA, Butt AK, Azhar M, Hanif M, Izhar M, Tatakis DN. Non-surgical periodontal therapy reduces coronary heart disease risk markers: a randomized controlled trial. J Clin Periodontol. 2012 Nov;39(11):1065-74. doi: 10.1111/j.1600-051X.2012.01942.x. Epub 2012 Sep 11. PMID 22966824

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 100 CHD patients recruited from Cardiology department of MY hospital, Indore, were evaluated at department of Periodontology, GDC Indore, for final selection.
Groups:
- Experimental: Periodontal intervention in the form of scaling and root planing by:
  1. ultrasonic piezoelectric scaler (frequency of 28-36 KHz) and
  2. gracey curets (set of 7 instruments number 1-14) to remove supra and subgingival calculus on teeth, is completed in two appointments of 45 to 60 min, within 24 hours
  piezoelectric ultrasonic scaler (frequency of 28-36 KHz): Periodontal treatment in the form of scaling and root planing (SRP) is provided to the patients assigned to the experimental group, after baseline examination. Scaling is performed using piezoelectric ultrasonic scaler (frequency of 28-36 KHz) and root planing is performed using area specific Gracey curettes (set of 7 instruments number #1-14). SRP is completed in two appointments of 45 min to 1 hour, within 24 hours period.
  Gracey curettes: set of 7 instruments number #1-14
Period: Overall Study
Arm/Group | Experimental | Control
Started | 35 | 35
Completed | 30 | 25
Not Completed | 5 | 10

BASELINE CHARACTERISTICS:
Population: All are CHD patients - never smoker, without any other systemic disease
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.43 (10.31) | 60.21 (9.23) | 60.30 (9.56)
Gender [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 23 | 26 | 49
Region of Enrollment [Number; unit: participants]
  India | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in C-Reactive Protein Level at 6 Months
Description: Change from baseline in high-sensitivity C-reactive protein level assessed quantitatively by immunoturbidimetric analysis at 6 months.
Time Frame: Baseline and 6 months
Population: All patients suffered from CHD and Periodontitis both.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mg/L | 6.30 (7.53) | 4.94 (2.04)

2. Secondary Outcome: Change From Baseline in C-Reactive Protein Level at 1 Month
Description: Change from baseline in high-sensitivity C-reactive protein level assessed quantitatively by immunoturbidimetric analysis at 1 month.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mg/L | 6.21 (1.92) | 4.31 (2.43)

3. Secondary Outcome: Change From Baseline in C-Reactive Protein Level at 3 Month
Description: Change from baseline in high-sensitivity C-reactive protein level assessed quantitatively by immunoturbidimetric analysis at 3 months.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mg/L | 6.22 (3.64) | 4.09 (1.82)

4. Secondary Outcome: Change From Baseline in Lipid Profile at 1 Month
Description: Change from baseline in lipid profile assessed at 1 month.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mg/dl | 35.67 (21.67) | 25.20 (6.48)

5. Secondary Outcome: Change From Baseline in Lipid Profile at 3 Months
Description: Change from baseline in lipid profile assessed at 3 months.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mg/dl | 33.70 (19.53) | 26.08 (7.14)

6. Secondary Outcome: Change From Baseline in Lipid Profile at 6 Months.
Description: Change from baseline in lipid profile assessed at 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mg/dl | 32.39 (18.43) | 26.24 (6.50)

7. Secondary Outcome: Change From Baseline WBC Profile at 1 Month
Description: Change from baseline in white blood cell profile assessed at 1 month.
Time Frame: Baseline and 1 month
Measure: Mean (Standard Deviation); unit: per cmm
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
per cmm | 8023.33 (2463.06) | 7448.00 (912.01)

8. Secondary Outcome: Change From Baseline WBC Profile at 3 Months
Description: Change from baseline in white blood cell profile assessed at 3 months.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: per cmm
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
per cmm | 7750 (1727.62) | 8260 (1830.76)

9. Secondary Outcome: Change From Baseline WBC Profile at 6 Months
Description: Change from baseline in white blood cell profile assessed at 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: per cmm
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
per cmm | 7553.33 (1634.91) | 8384.00 (1171.07)

10. Secondary Outcome: Systolic Blood Pressure at 1 Month
Description: Systolic blood pressure at 1 month.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mmHg | 130.00 (19.69) | 120.56 (17.60)

11. Secondary Outcome: Systolic Blood Pressure at 3 Months
Description: Systolic blood pressure at 3 months.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mmHg | 125.47 (16.27) | 118.56 (14.23)

12. Secondary Outcome: Systolic Blood Pressure at 6 Months
Description: Systolic blood pressure at 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mmHg | 123.70 (15.72) | 120.88 (14.56)

13. Secondary Outcome: Change From Baseline Periodontal Parameter- Periodontal Probing Depth at 6 Months
Description: Change from baseline in periodontal parameter- periodontal probing depth at 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mm | 1.78 (0.54) | 1.86 (0.31)

14. Secondary Outcome: Change From Baseline Periodontal Parameter- Gingival Index at 6 Months
Description: Change from baseline in periodontal parameter- gingival index at 6 months. Scale ranges for Total Gingival Index - Minimum score (0) and maximum score (3).
  Score 0 represents better outcome and higher scores represent worst outcome. Score per person are calculated by taking average of scores for 6 sites of all teeth recorded.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
Scores on a scale | 0.49 (0.19) | 1.32 (0.13)

15. Secondary Outcome: Change From Baseline Periodontal Parameter- Plaque Index at 6 Months
Description: Change from baseline in periodontal parameter- plaque index at 6 months. Scale ranges for Total Plaque Index - Minimum score (0) and maximum score (3). Score 0 represents better outcome and higher scores represent worst outcome. Score per person are calculated by taking average of scores for 6 sites of all teeth recorded.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
Scores on a scale | 0.80 (0.62) | 1.15 (0.14)

16. Secondary Outcome: Change From Baseline Periodontal Parameter- Bleeding on Probing at 6 Months
Description: Change from baseline in periodontal parameter- bleeding on probing at 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: percentage of sites
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
percentage of sites | 38.97 (12.93) | 83.20 (13.02)

17. Secondary Outcome: Change From Baseline Periodontal Parameter- Clinical Attachment Loss at 6 Months
Description: Change from baseline in periodontal parameter- clinical attachment loss at 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mm | 2.85 (0.59) | 2.78 (0.64)

18. Secondary Outcome: Diastolic Blood Pressure at 1 Month
Description: Diastolic blood pressure at 1 month.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mmHg | 83.87 (10.51) | 76 (9.98)

19. Secondary Outcome: Diastolic Blood Pressure at 3 Months
Description: Diastolic blood pressure at 3 months.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mmHg | 80.67 (9.66) | 76.48 (7.90)

20. Secondary Outcome: Diastolic Blood Pressure at 6 Months
Description: Diastolic blood pressure at 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Experimental | Control
Number analyzed (Participants) | 35 | 35
mmHg | 80.07 (9.12) | 76.64 (7.78)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were not collected
Arm/Group | Experimental | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
populations were taken only from a single center, the dropout, strict inclusion criteria, total number of patients to be included in the study was limited, influence of medical drug management of CHD not taken into consideration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No